CLINICAL TRIAL: NCT06647914
Title: Predicting Disease Progression in Atrial Fibrillation: A Multiparametric Approach for Prognostic Marker Identification and Personalized Patient Management
Acronym: PAMP FA
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Collaborators: Federico II University (Other); Irccs Sdn (Other); Marche Polytechnic university, Ancona, Italy (Unknown)
Responsible Party: Sponsor
Other Study IDs: PNRR-MCNT2-2023-12378472
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-09

CONDITIONS: Atrial Fibrillation (AF)
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project leverages artificial intelligence (AI) to decipher Atrial Fibrillation (AF) progression and optimize treatment strategies. By recruiting a diverse cohort of 322 AF patients, we will gather a robust multiparametric dataset including clinical, genetic, electrocardiographic, and echocardiographic data. Harnessing AI, we will extract and correlate hidden components within ECG-obtained P-wave data and echocardiographic studies with atrial fibrosis, culminating in an atrial fibrosis score (AFS). The AFS will non-invasively predict fibrosis extent and AF clinical progression, including metrics like rehospitalization, cardiac morbidity, and mortality. Ultimately, this endeavor aims to improve AF patient management, significantly reducing healthcare costs, and enhancing patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

* History of paroxysmal or persistent atrial fibrillation
* Clinical indication for Atrial Fibrosis (AF) ablation according to the 2020 ESC Guidelines

Exclusion Criteria:

* Age below 18 years old
* Refusal to sign consent
* Noncompliance with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited at the two Clinical Institution of I.R.C.C.S. Policlinico San Donato and Federico II University of Naples, with the same study protocol approved by the Institutional Board of the respective Institution.
Sampling Method: Probability Sample
Enrollment: 322 (Estimated)
Dates: Start 2025-09-03 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
A composite clinical point used to evaluate the Atrial Fibrosis Score prognostic capability | Partecipants will be assessed at the baseline and at 6 months and 12 months time points. The AFS Prediction Model Testing will start at 9 months after the beginning of the patients enrollment.
  The clinical endpoint will be composed by rehospitalization, cardiac morbidity and total mortality data